CLINICAL TRIAL: NCT00063206
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Study of a Flexible Dose of DVS-233 SR in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 in Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 3151A1-304
Record Dates: First submitted 2003-06-23; First posted 2003-06-25 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
Keywords: Depressive Disorder, Major; Depression, Involutional
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
Primary: To compare the antidepressant efficacy and safety of subjects receiving DVS-233 SR versus subjects receiving placebo.

Secondary: To assess the response of subjects receiving DVS-233 SR for the clinical global evaluation, functionality, general well-being, pain, and remission (Hamilton Psychiatric Rating Scale for Depression, 17-item [HAM-D<sub>17</sub>] < 7) versus those subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a primary diagnosis of major depressive disorder (MDD)
* Depressive symptoms for at least 30 days prior to the screening visit
* Minimum screening and study day -1 (baseline) scores of 20 on the Hamilton Psychiatric Rating Scale for Depression (HAM D<sub>17</sub>)

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past
* Treatment with venlafaxine (immediate release [IR] or extended release [ER]) within 90 days of study day 1
* Known hypersensitivity to venlafaxine (IR or ER)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Liebowitz MR, Yeung PP, Entsuah R. A randomized, double-blind, placebo-controlled trial of desvenlafaxine succinate in adult outpatients with major depressive disorder. J Clin Psychiatry. 2007 Nov;68(11):1663-72. doi: 10.4088/jcp.v68n1105. PMID 18052559